CLINICAL TRIAL: NCT04962035
Title: Neurocognitive Scores of Predominantly Formula Fed Preterm Infants in Early Childhood Years
Brief Title: Neurocognitive Follow-Up (FU) Study
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 2006INF
Record Dates: First submitted 2021-04-29; First posted 2021-07-14 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Developmental Delay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alprem RTF Brain Follow-up: Neurocognitive Follow-up of children previously having participated in the Alprem RTF study
  Interventions: Other: Neurocognitive Follow-up

INTERVENTIONS:
Other: Neurocognitive Follow-up — Standard clinical and parent-reported outcomes on cognitive development, temperament and overall health conditions.

SUMMARY:
This is a follow-up study of a recently completed trial (17.14.INF) evaluating the growth of pre-term infants. Enrolled children will undergo neurocognitive assessments at 18- and 24-months of corrected age (CA).

DETAILED DESCRIPTION:
This is a follow-up study of a recently completed multi-center, prospective, single-arm, open-label interventional trial (17.14.INF - Alprem RTF: NCT03728764) evaluating the growth of pre-term infants receiving a two-stage PTF feeding system while in the neonatal care unit and continuing until 30 days post-discharge.

Enrolled children will undergo neurocognitive assessments at 18- and 24-months of corrected age (CA). The timing of the cognitive assessments aligns with routine check-up visits and reflect the period at which developmental delays may first become evident.

ELIGIBILITY:
Inclusion Criteria:

1. Infants / children born prematurely who were enrolled into the original clinical trial and who are less than 24 m of CA.
2. Having obtained his / her parents' (or his or her legally accepted guardian written informed consent and having evidence of personally signed and dated informed consent document indicating that the child's parent(s) / legal guardian has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Infants identified retrospectively as not meeting the inclusion or exclusion criteria for the original study.

Ages: 17 Months to 25 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants who have previously participated in the 17.14.INF Alprem RTF study are eligible to participate, wherein preterm infants of gestational age ≥ 27 weeks and ≤ 32 weeks with body weight <1500g and appropriate for gestational age (AGA) as defined by weight ≥10 percentile and ≤90 percentile on the Fenton growth chart had been enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Bayley-III scores at 24 months | 24 months of CA
  Bayley Scales of Infant and Toddler Development, third edition (Bayley-III) cognitive score at 24 months of corrected age (CA). Composite scores range 40-160, with a mean of 100 and SD of 10 points. A composite score of 70 or less is an indication of a delay in child neurocognitive development.

SECONDARY OUTCOMES:
Bayley-III scores at 18 months | 18 months of CA
  Bayley Scales of Infant and Toddler Development, third edition (Bayley-III) cognitive score at 18 months of corrected age (CA). Composite scores range 40-160, with a mean of 100 and SD of 10 points. A composite score of 70 or less is an indication of a delay in child neurocognitive development.
Weight | At enrollment, 18 and 24 months of CA
  Child weight (g)
Length/height | At enrollment, 18 and 24 months of CA
  Child length/height (cm)
Head circumference | At enrollment, 18 and 24 months of CA
  Child head circumference (cm)
Child temperament scores | At 18 and 24 months of CA
  Parent-reported child temperament questionnaire validated specifically for children between the ages of 18 and 36 months
Developmental Milestone scores | At 18 and 24 months of CA
  Parent-reported achievements of specific age-appropriate milestones (yes/no responses to child performing specific milestones or not)
Number of healthcare usage | At 18 and 24 months of CA
  Retrospective parent-reported recall of the number of healthcare usage and hospitalizations
Feeding patterns | At 18 and 24 months of CA
  Feeding practice outcomes collected retrospectively at each visit via a parent-reported questionnaire related to breastfeeding duration, prevalence of formula feeding, and age at initiation of complementary feeding

CONTACTS AND LOCATIONS:
Locations (3):
- Klinika Chorob Dzieci, Uniwersytecki Szpital Dzieciecy, Krakow, Poland
- Slovakia (2):
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwinta P, Lazarova S, Demova K, Chen Y, Hartweg M, Krattinger LF, Fumero C, Buczynska A, Durlak W, Uhrikova Z, Kozar M, Samuel TM, Zibolen M. Effects of two-stage preterm formulas on growth, nutritional biomarkers, and neurodevelopment in preterm infants. Front Pediatr. 2024 Nov 22;12:1427050. doi: 10.3389/fped.2024.1427050. eCollection 2024. PMID 39649400